CLINICAL TRIAL: NCT01835886
Title: Study to Assess if Ability to Ascend and Descend Stairs Within 30 Seconds Will Prove to be a Reliable and Valid Outcome Measure in Individuals With Pulmonary Disease
Brief Title: Study to Assess Stairs as an Outcome Measure in Individuals With Pulmonary Disease
Acronym: TSCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 183-12
Record Dates: First submitted 2013-04-01; First posted 2013-04-19 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Pulmonary Disease
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Performs stair-climbing (Experimental): Performs stair climbing
  Interventions: Other: Patients will ascend and descend a flight of 10 steps

INTERVENTIONS:
Other: Patients will ascend and descend a flight of 10 steps — Patients referred to pulmonary rehabilitation with documented lung disease will ascend and descend a flight of 10 steps for a period of 30 seconds

SUMMARY:
To determine if stair climbing can be used as a measure of progress in persons with pulmonary disease.

DETAILED DESCRIPTION:
Protocol Title: The Reliability and Validity of the Timed Stair Climbing Test (TSCT) as an Outcome Measure in Individuals with Pulmonary Disease.

Background An important part of pulmonary rehabilitation is the ability to document progress. Commonly used outcome measures include walking tests like the Six Minute Walk Test (6MWT) and the Shuttle Walk Test, MET levels and questionnaires. A recent study by Annegarn1 et al., analyzed responses from 820 Chronic Obstructive Pulmonary Disease (COPD) patients. While 35% of respondents cited stair climbing as a problematic Activity of Daily Living (ADL), there are very few studies looking at stair climbing ability as an outcome measure.

Step tests using a riser and metronome have long been used as a fitness measure for healthy subjects but can be challenging to administer to a non healthy population and do not mimic the challenge of actually mounting a series of steps. Many of the existing stair climbing studies which use actual stairs for testing are distance based and examine stair climbing as a predictor for outcomes following lung surgery. One study conducted by Randolph2 et al., attempted to compare stair climbing ability and Pulmonary Function Tests (PFTs) as predictors of post-thoracotomy outcomes. Brunelli3 et al., looked at stair climbing as a useful predictor of cardiopulmonary complications following lung resection. Both studies concluded that the stair climbing test was clinically useful.

Bean4 developed a stair climbing test called the Stair Climb Power Test that incorporated an element of time by asking subjects to climb a staircase of ten stairs as quickly and safely as possible and looked at the relationship between muscle strength and functional performance.

The Six Minute Walk Test is well established as a valid and reliable outcome measure for this population5. A study by Dreher6 et al., in 2008 attempted to compare a stair climbing test with the Six Minute Walk Test. Using a randomized cross-over design, they looked at sixteen COPD patients and found that pathophysiological changes during a six minute walk test did not anticipate changes found during stair climbing in patients with severe COPD.

All of this points to the fact that a timed stair climbing test has the potential to serve as a unique and valuable outcome measure for patients with respiratory compromise. It is well understood that many people with pulmonary disease, especially those who live in urban areas, unavoidably encounter stairs. While the six minute walk test requires at minimum a long straight hallway with a hard surface for administration7 even that is not always readily available. The Timed Stair Climbing Test could provide an outcome measure that is easily administered and could be utilized in outpatient and inpatient settings as well as in the home environment.

Questions Addressed Is the Timed Stair Climbing Test a reliable and valid measure to use to assess endurance in individuals with pulmonary disease when compared to 6MWT?

Research Design Methodological Research design to establish validity and reliability of the Timed Stair Climbing Test will be used. Test scores from 6MWT and TSCT will be compared, using patients with documented pulmonary disease who participate in pulmonary rehabilitation. All testing will take place on the premises of The Alice Lawrence Center for Health and Rehabilitation located on the third floor of the Linsky Building, Petrie Campus of Beth Israel Medical Center at First Ave and 16th Street in New York City. Screening of subjects and test administration will be conducted by investigators and will be limited to staff members who are licensed Physical Therapists or Exercise Physiologists with ACLS certification operating under the supervision of Dr. Jonathan Raskin, MD, director of the center.

Administration of the 6MWT is currently part of the usual standard of care for pulmonary rehabilitation patients attending the center. It is performed twice, one on evaluation and once later towards the end of a person's series of sessions. American Thoracic Society guidelines for administering the 6MWT will be followed.

The Timed Stair Climbing Test will be added to subject's initial evaluations and discharge sessions for research purposes. For the TSCT patients will be supervised while ascending and descending a flight of 10 steps with 7 inch risers for 30 seconds as timed by a stop watch. Number of steps achieved, oxygen saturation, rate of perceived exertion, dyspnea, heart rate and use or non-use of a hand rail will be recorded. Vital signs will be continuously monitored. As with the 6MWT, subjects will be allowed to use supplemental oxygen if it has been prescribed for them. Whether the test was performed on room air or with supplemental oxygen will be recorded in the test results. Oxygen delivery system and level of oxygen flow and how equipment was managed will also be recorded in the test results. Subjects will have the option of relying on any assistive devices to which they are accustomed and use or non use of canes, handrails, orthoses etc will be recorded.

Subjects will be deemed fit to attempt the stair climbing task by the investigators only if they are in no apparent distress, have a resting heart rate above 50 and below 120, resting blood pressure above 90/50 and below 150/90 and no complaints of pain or dyspnea greater than 2/10 at rest and an oxygen saturation level greater than 90% at rest as measured by pulse oximeter. The test will be terminated after 30 seconds or in the event of complaints of pain or dyspnea greater than 4/10, an increase in heart rate greater than 40 beats over resting or a decrease in oxygen saturation to below 86% or at any time at the request of the patient.

Inclusion Criteria: This study will include patients with documented pulmonary disease who underwent a course of pulmonary rehabilitation at The Alice Lawrence Center for Health and Rehabilitation consisting of 10 or more sessions.

Exclusion Criteria: The following will be excluded from the study:

1. Patients who are unable to perform a follow-up 6MWT or TSCT or who are lost to follow-up.
2. Patients who have orthopedic or neurological conditions (significant limitations in ambulation or stair climbing) that limit participation in pulmonary rehabilitation.

Data Analysis Pearson-Product Moment Correlation Coefficient or Spearman Rho for Convergent Validity will be used to compare 6MWT and TSCT results. Intra-class Correlation Coefficient for Intra-rater, Inter-rater, and Test-retest Reliability will also be computed.

Dr. David Lucido was consulted for his expertise as a biostatistician. He suggested that 30 to 60 participants would be an adequate sample size for purposes of the study.

Significance This study would help to determine if the Timed Stair Climbing Test is a useful outcome measure for people with pulmonary disease.

References

1. Annegarn J, Meijer K, Passos VL, Stute K, Wiechert J, Savelberg HH, Schols AM, Wouters EF, Spruit MA; Ciro+ Rehabilitation NetworkJ Am Med Dir Assoc. Problematic activities of daily life are weakly associated with clinical characteristics in COPD. 2012 Mar;13(3):284-90. Epub 2011 Feb 17.
2. Bolton JW, Weiman DS, Haynes JL, Hornung CA, Olsen GN, Almond CH. Stair climbing as an indicator of pulmonary function. Chest. 1987 Nov;92(5):783-8.
3. Brunelli A, Refai MA, Monteverde M, Borri A, Salati M, Fianchini A: Stair climbing test predicts cardiopulmonary complications after lung resection. Chest 2002;121:1106-1110.
4. Bean, JF, Kiely DK, LaRose S,et al. Is stair climb power a clinically relevant measure of leg power impairments in at-risk older adults? Arch Phys Med Rehabil. 2007:88:604-609.
5. Robert A Wise and Cynthia D Brown Minimal Clinically Important Differences in the Six-Minute Walk Test and the Incremental Shuttle Walking Test COPD: Journal of Chronic Obstructive Pulmonary Disease, 2005, Vol. 2, No. 1 : Pages 125-129.
6. Dreher M, Walterspacher S, Sonntag F, Prettin S, et al. (2008). Exercise in severe COPD: is walking different from stair-climbing? Respiratory Medicine 102(6):912-8.
7. American Thoracic Society Statement (2002) Guidelines for the Six-Minute Walk Test Am J Respir Crit Care Med Vol 166. pp 111-117.

ELIGIBILITY:
Inclusion Criteria:

* This study population will consist of patients with documented pulmonary disease who underwent a course of pulmonary rehabilitation at The Alice Lawrence Center for Health and Rehabilitation consisting of 10 or more sessions

Exclusion Criteria:

* Patients who have orthopedic or neurological conditions (significant limitations in ambulation or stair climbing) that limit participation in pulmonary rehabilitation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Timed Stair Climbing Test Assessing Change Between Initiation and at Completion of Pulmonary Rehabilitation Sessions | Ascent and descent of stairs will be assessed prior to initiating and following 18 to 36 weeks of outpatient pulmonary rehabilitation
  Subjects will be asked to ascend and descend a flight of 10 steps both at initiation and completion of a course of pulmonary rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Ted L Marks, DPT, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center, New York, New York, United States